CLINICAL TRIAL: NCT02167048
Title: Effects of Low-dose Versus Normal-dose Psychostimulants on Executive Functions in Individuals With Attention-Deficit Hyperactivity Disorder
Brief Title: Low-dose vs. Normal-dose Psychostimulants on Executive Functions in Individuals With ADHD
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Adele Diamond, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H14-00224
Record Dates: First submitted 2014-06-11; First posted 2014-06-18 (Estimated); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Attention Deficit Hyperactivity Disorders
Keywords: Attention Deficit Hyperactivity Disorders; Executive Function; Methylphenidate; Psychostimulants; Adolescent; Child; Working Memory; Prefrontal Cortex; Attention; Cognitive Function; Inhibition
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Inhibition, Psychological

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Normal-dose Psychostimulant, Low-dose (Experimental): Normal-dose: Dose participants are currently taking as part of their prescription (on more than or equals to 20 mg/day of Psychostimulants) Low-dose: Half the normal dose
  Interventions: Drug: Psychostimulants
- Low-dose Psychostimulants, Normal-dose (Active Comparator): Normal-dose: Dose participants are currently taking as part of their prescription (on more than or equals to 20 mg/day of Psychostimulants) Low-dose: Half the normal dose
  Interventions: Drug: Psychostimulants
- No intervention, No intervention (No Intervention): This arm is completely no intervention, and is ONLY for healthy volunteers. We are testing healthy volunteers of the same age to give us an estimate of order effects to help us correct for better performance in the 2nd session due simply to taking the same tests twice (note: the tests are Version A and B).

INTERVENTIONS:
Drug: Psychostimulants — Participants will be tested twice 2 weeks apart. All will continue on their normal Psychostimulant dose up until 3 days before the testing day. 3 days before their 1st testing session, half the participants will start on either their current-dose of Psychostimulant or half their current dose depending on the arm they were randomized to (we provide those pills).
  To control for different pharmacokinetics of the Psychostimulant medications, a given participant will be tested at roughly the peak time for his/her specific version of Psychostimulant and at the same time of day for his/her two testing sessions.
  Arms: Low-dose Psychostimulants, Normal-dose; Normal-dose Psychostimulant, Low-dose

SUMMARY:
This double-blind crossover study aims to compare cognitive performance (e.g., working memory, selective attention and cognitive flexibility) of children ages 6-18 years diagnosed with ADHD of the combined type (ADHD-C) or inattentive-type (ADHD-IA) and currently on > 20 mg/day of psychostimulants (psychostimulants) on: a) their current dose of psychostimulants, vs. b) a lower-dose of psychostimulants (half of their current dose).

The investigators hypothesize that the lower-dose psychostimulants will result in better cognitive performance than moderate-to-high doses of psychostimulants.

DETAILED DESCRIPTION:
Attention-deficit hyperactivity disorder (ADHD) is a neurodevelopmental disorder characterized by attention deficits, hyperactivity, or impulsive actions that are not appropriate for the individuals' age (Barkley 1997). These behavioural issues arise relatively early in life, typically before the age of 12, and continue to persist into adulthood in many cases (Barkley 1997). In school-aged children, ADHD is associated with low academic achievement, poor school performance, anxiety and depression.

Symptoms are divided into inattention (e.g., easily distracted, difficulty focusing on & completing a task), hyperactivity (e.g., constantly in motion, fidgets, squirms, talks non-stop), and impulsivity (e.g., difficult waiting one's turn, interrupting others). Three subtypes of ADHD have been identified: predominantly inattentive (ADHD-I), predominantly hyperactive-impulsive (ADHD-H), and the combined type (ADHD-C).

Psychostimulants in medium to high doses acts to inhibit re-uptake of dopamine by the dopamine transporter (DAT), resulting in increased dopamine concentrations in the synapse. DAT is abundant in the striatum, which is implicated in hyperactivity and impulsivity aspects of ADHD. However, DAT is sparse in prefrontal cortex (PFC), which plays a critical role in subserving executive functions. Executive functions (EFs; also called cognitive control or self-regulation) are a group of processes involved in concentration, focused attention, self-control, cognitive flexibility, problem-solving, and working memory (refs: Diamond, 2013; Jacques & Marcovitch, 2010). Thus the number of high risk alleles of the gene that codes for the dopamine transporter (DAT1) are associated with hyperactivity (which depends on the striatum) but not inattention or EF deficits (which depend on PFC; refs: Jucaite et al., 2005; Waldman et al., 1998.

The action of low doses of psychostimulants has been shown to be different, however. At low doses psychostimulants has been demonstrated to act preferentially on PFC, increasing dopamine release (refs: Berridge et al., 2006; Schmeichel & Berridge, 2013; Spencer et al, 2012). Thus, moderate to high doses of psychostimulants (doses most often prescribed for children and youths with ADHD) probably do not improve PFC function or EFs, or worse, may actually impair cognitive function, leaving a patient feeling more in a daze.

Optimal dosing for psychostimulants in children and youths with ADHD is usually determined by parents' reports of improved behaviour, almost never by performance on cognitive measures. We propose to look at cognitive performance on measures of attention, working memory, planning, etc. in children and youths with ADHD on their current dose of psychostimulants and on half that much (order counterbalanced across participants).

Purpose/Objectives: This double-blind crossover study aims to compare cognitive performance (e.g., working memory, selective attention and cognitive flexibility) of children ages 6-18 years diagnosed with ADHD of the combined type (ADHD-C) or inattentive-type (ADHD-IA) and currently on > 20 mg/day of psychostimulants on their current dose of psychostimulants and on a lower-dose of psychostimulants (half of their current dose), order counterbalanced across subjects.

To give us an estimate of order effects to help us correct for better performance in the 2nd session due simply to taking the same cognitive tests twice (note: the tests are Version A and B), we will also be recruiting healthy volunteers to serve as a control group. This control group will be strictly no intervention.

Hypotheses: The investigators hypothesize that lower-dose psychostimulants will result in better cognitive performance than moderate-to-high doses of psychostimulants.

ELIGIBILITY:
Inclusion Criteria:

* Between the chronological ages of 6 and 18 years
* Average to above-average IQ (Parental report of an IQ above 90; we will take their word for it)
* Meet DSM-V criteria for ADHD (Combined type or Inattentive type)
* Currently treated with and responding to oral Psychostimulants >= 20 mg/day and not on a "drug holiday"
* Stable on current Psychostimulant dose for at least 2 weeks
* Able to communicate (understand, speak, and write) in English without the aid of an interpreter
* Able to execute simple manual response (button-press) as required for our tasks
* The child and parent give assent and consent respectively for the child's participation in this study

Exclusion Criteria:

* Patients with significant prior or current medical conditions that could impact neuropsychological performance such as traumatic brain injury, hypoxia, or unstable diabetes.
* Have any medical condition that could markedly increase sympathetic nervous system activity (e.g. catecholamine-secreting neural tumor), or who are taking a medication on a daily basis (e.g. pseudoephedrine, oral steroids) that has sympathomimetic activity. Note: regular on-label use of inhalers for asthma (e.g., albuterol, steroidal) is permitted
* Taking any psychotropic medication other than on-label Psychostimulants specifically prescribed to treat ADHD
* Have a major, uncorrected sensory impairment (e.g. significant hearing impairment despite hearing aids)
* Lack sufficient English language skills to perform our tasks
* Are taking medications other than their specifically prescribed Psychostimulants that may affect cognitive skills
* Have a documented history of Dyslexia (this may skew results on our cognitive measures), Bipolar I or II, psychosis, Depression, Autism Spectrum Disorders, or Disruptive Mood Dysregulation Disorder
* Have a past history of any severe adverse reaction to lowering of Psychostiumlant dose
* Patient has been non-compliant with Psychostimulants or is on a "drug holiday"
* Parental report of an IQ below 90 (we will take their word for it)

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 52 (Estimated)
Dates: Start 2014-06; Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Executive Functions (difference in performance on the two Psychostimulants doses) | Day 1
  Executive Functions consist of selective attention, working memory, response inhibition, reasoning, and set switching. Each of those component abilities will be assessed, scores converted to z scores, and a composite score assigned to each subject for each test session.
Executive Functions (difference in performance on the two Psychostimulant doses) | 2 weeks
  Executive Functions consist of selective attention, working memory, response inhibition, reasoning, and set switching. Each of those component abilities will be assessed, scores converted to z scores, and a composite score assigned to each subject for each test session.

CONTACTS AND LOCATIONS:
Overall Officials: Adele Diamond, Ph.D., Principal Investigator — Department of Psychiatry, University of British Columbia
Locations (1):
- Developmental Cognitive Neuroscience Lab, Department of Psychiatry, University of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Barkley RA. Behavioral inhibition, sustained attention, and executive functions: constructing a unifying theory of ADHD. Psychol Bull. 1997 Jan;121(1):65-94. doi: 10.1037/0033-2909.121.1.65. PMID 9000892
- [Background] Diamond A. Executive functions. Annu Rev Psychol. 2013;64:135-68. doi: 10.1146/annurev-psych-113011-143750. Epub 2012 Sep 27. PMID 23020641
- [Background] Jacques, S., & Marcovitch, S. (2010). Development of executive function across the life span. In W. F. Overton (Ed.), Cognition, biology and methods across the lifespan: Volume 1 of the handbook of life-span development (pp. 431-466). Hoboken, NJ: Wiley.
- [Background] Jucaite A, Fernell E, Halldin C, Forssberg H, Farde L. Reduced midbrain dopamine transporter binding in male adolescents with attention-deficit/hyperactivity disorder: association between striatal dopamine markers and motor hyperactivity. Biol Psychiatry. 2005 Feb 1;57(3):229-38. doi: 10.1016/j.biopsych.2004.11.009. PMID 15691523
- [Background] Waldman ID, Rowe DC, Abramowitz A, Kozel ST, Mohr JH, Sherman SL, Cleveland HH, Sanders ML, Gard JM, Stever C. Association and linkage of the dopamine transporter gene and attention-deficit hyperactivity disorder in children: heterogeneity owing to diagnostic subtype and severity. Am J Hum Genet. 1998 Dec;63(6):1767-76. doi: 10.1086/302132. PMID 9837830
- [Background] Berridge CW, Devilbiss DM, Andrzejewski ME, Arnsten AF, Kelley AE, Schmeichel B, Hamilton C, Spencer RC. Methylphenidate preferentially increases catecholamine neurotransmission within the prefrontal cortex at low doses that enhance cognitive function. Biol Psychiatry. 2006 Nov 15;60(10):1111-20. doi: 10.1016/j.biopsych.2006.04.022. Epub 2006 Jun 23. PMID 16806100
- [Background] Schmeichel BE, Berridge CW. Neurocircuitry underlying the preferential sensitivity of prefrontal catecholamines to low-dose psychostimulants. Neuropsychopharmacology. 2013 May;38(6):1078-84. doi: 10.1038/npp.2013.6. Epub 2013 Feb 6. PMID 23303075
- [Background] Spencer RC, Klein RM, Berridge CW. Psychostimulants act within the prefrontal cortex to improve cognitive function. Biol Psychiatry. 2012 Aug 1;72(3):221-7. doi: 10.1016/j.biopsych.2011.12.002. Epub 2011 Dec 29. PMID 22209638